CLINICAL TRIAL: NCT04107454
Title: Effect of Treatment With the Ablative Fractional Carbodioxide Laser in Vulvar Lichen Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Deka Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VLS-AFCL
Record Dates: First submitted 2019-09-24; First posted 2019-09-27 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Lichen Sclerosus Et Atrophicus of the Vulva
Keywords: Lichen sclerosus
MeSH Terms: conditions — Lichen Sclerosus et Atrophicus

STUDY DESIGN:
Intervention Model Description: The study is designed as a randomized placebo-controlled study
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active group (Active Comparator): The laser setting is: Power 24 W, exposure time 400 microsec, density 6,4 %, pulse energy 23,2 mJ, fluenz 1,18J/cm2, emission mode DP, DOZ Dwell 400, DOT spacing 1000.
  Interventions: Device: Active microablative fractional CO2 laser designed as SmartXide Touch C60, CO2 laser system for MonaLisa Touch, DEKA, Florence
- Placebo group (Placebo Comparator): Laser setting is a sham dose:power 0, 5 W, exposure time 400 microsec, DOT spacing 1000
  Interventions: Device: Sham microablative fractional CO2 laser designed as SmartXide Touch C60, CO2 laser system for MonaLisa Touch, DEKA, Florence

INTERVENTIONS:
Device: Active microablative fractional CO2 laser designed as SmartXide Touch C60, CO2 laser system for MonaLisa Touch, DEKA, Florence — Active application of laser radiation on the vulvar skin. The laser setting is: Power 24 W, exposure time 400 microsec, density 6,4 %, pulse energy 23,2 mJ, fluenz 1,18J/cm2, emission mode DP, DOZ Dwell 400, DOT spacing 1000.
  Arms: Active group
Device: Sham microablative fractional CO2 laser designed as SmartXide Touch C60, CO2 laser system for MonaLisa Touch, DEKA, Florence — Sham application of laser radiation on the vulvar skin. Laser setting is a sham dose:power 0, 5 W, exposure time 400 microsec, DOT spacing 1000
  Arms: Placebo group

SUMMARY:
Aim of this study is to evaluate the therapeutic effect of the laser treatment in vulvar LS, mainly the reduction of existing symptoms. As measured by visual analogue scale (VAS) symptoms as itching, burning, pain will be determined six weeks after the last laser treatment. Secondary endpoints will be sexual function measured with the female sexual function index (FSFI) and the vulvar skin changes measured by the Lichen score (LS).

Regular photo-documentation of the treated skin will demonstrate a potential change of the tissue.

DETAILED DESCRIPTION:
Lichen sclerosus (LS) is a vulvar dermatosis that changes the skin to white plaques (lichenification), less elasticity (sclerosis) and the tissue shows contractions with erosions and fissures. Gold standard for the therapy of LS is the topical application of ultrapotent corticosteroids, proper treatment reverses the underlying inflammation of LS, reduces symptoms as itching and burning and may lower the risk of getting vulvar cancer. While useful, steroid creams may have serious side effects that include thinning of the skin, fungal infections, and lowering the immune system. Treatment with the fractional microablative carbodioxide Laser is a minimal invasive procedure. In the literature only few published reliable data in laser therapy of vulvar skin diseases can be found, there is only one survey especially for the treatment of vulvar LS. However, published data show a potential that justifies the use of this method for the indication in treating LS.

Aim of this study is to evaluate the therapeutic effect of the laser treatment in vulvar LS, mainly the reduction of existing symptoms. But there is little comparable data, so the necessary frequency of treatment, the dose of laser application, additional use of corticosteroid or the sustainability is not yet known

Aim of this study is to evaluate the therapeutic effect of the laser treatment in vulvar LS, mainly the reduction of existing symptoms. As measured by visual analogue scale (VAS) symptoms as itching, burning, pain will be determined six weeks after the last laser treatment. Secondary endpoints will be sexual function measured with the female sexual function index (FSFI) and the vulvar skin changes measured by the Lichen score (LS).

Regular photo-documentation of the treated skin will demonstrate a potential change of the tissue.

Primary endpoint will be the outcome after laser application, the change in symptoms between both groups. As secondary endpoint it is important to see, weather sexual functions will be influenced in this therapy.

The study is designed as a randomized placebo-controlled study.

Inclusion criteria: All patients are treated in the dysplasia unit of the university gynecological hospital of Bern. They have a histological confirmation of LS or a clinical diagnosis of LS according to the lichen-score. Informed consent will be oral and written. The minimum age is 18 years

Exclusion criteria: Pregnancy, local bacterial or parasitical infection, others severe dermatosis, Lichen-score < 5, vulvar cancer

All women who qualify for the study and signed informed consent will be grouped by computer-controlled randomization. All of them are informed, that they have to take part in three sequent sessions of treatment in the interval of three weeks and the defined follow -ups after six and twelve weeks.

The session starts with the application of an ointment for a local anesthesia in the vulvar region. Meanwhile they will answer the questionnaires (VAS for recording the vulvar symptoms, FSFI for the documentation of the sexual function, another questionnaire to evaluate the present situation).

After about 20 minutes the gynecologist will start the examination with a photo documentation of the vulva, then the laser application of the vulva is following. After the treatment a cream of silversulfadiazine (Flammazine) will be applied.

All personal data of the patients will be anonymized. The study specific intervention is an application of laser radiation on the vulvar skin.

The used laser instrument for this specific intervention is a microablative fractional CO2 laser designed as SmartXide Touch C60, CO2 laser system for MonaLisa Touch, DEKA, Florence. For the vulvar use the Hi-Scan V2LR scanning system has to be connected.

The laser setting is: Power 24 W, exposure time 400 microsec, density 6,4 %, pulse energy 23,2 mJ, fluenz 1,18J/cm2, emission mode DP, DOZ Dwell 400, DOT spacing 1000.

Projected are three sequent sessions in three weeks intervals. Application time takes approximately five minutes for the whole vulvar skin.

The study will compare two groups of patients, both fulfil the same criteria as a histological confirmation of LS or a clinical diagnosis of LS according to the lichen-score. They will be grouped by computer-controlled randomization in an active group and in a placebo group.

The active group will be treated by radiation with a real dose: power 24 W, exposure time 400 microsec, DOT spacing 1000.

The placebo group will be treated with a sham dose: power 0, 5 W, exposure time 400 microsec, DOT spacing 1000.

Both groups undergo the same procedures, they will have the same application time and application area. Except of the different radiation dose they undergo the same regimen.

ELIGIBILITY:
Inclusion Criteria:

* Women aged >18 years
* Women with histological assured or clinical confirmed Lichen sclerosus (Lichen score > 5)
* Informed Consent as documented by signature (Appendix Informed Consent Form)

Exclusion Criteria:

* Unable to read or understand study patient information document
* Patients with a legal guardian
* Refusal to participate
* Missing signed consent
* Pregnancy and lactation
* Proven bacterial or parasitic infection (clinical examination and/or vaginal wet mount)
* Vulvar cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Study enrollment possible for all participants with vulvar lichen sclerosus
Enrollment: 64 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Vulvar pain measured with the visual analog scale with a range from 0 (no pain, best Outcome) to 10(worst pain, worst Outcome) | End 12/2020. The measurements will be taken before each treatment and at the Follow-ups at 12 weeks and 18 weeks
  Primary objective of this study is the number of patients with reduction or cure of the symptoms of LS as itching, burning and vulvar pain after treatment is reduced. The effect will be measured with the visual analog scale.

SECONDARY OUTCOMES:
Sexual functioning measured with the Female Sexual Function Index (FSFI), each question ranges from 0 to 5 and the full scale score will be calculated(ranges from 2 (worst Outcome) to 36 (best Outcome)) | End 12/2020. The measurements will be taken before each treatment and at the Follow-ups at 12 weeks and 18 weeks
  Secondary objective is the awareness that the laser treatment leads to an improvement of the sexual function, e.g. amelioration the dyspareunia.he effect will be measured with the Questionaire FSFI.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Knabben, Dr. med., Principal Investigator — Inselspital Frauenklinik
Locations (1):
- Inselspital Frauenklinik, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No